CLINICAL TRIAL: NCT00322283
Title: Efficacy and Safety of Oglemilast in the Prevention of Exercise-Induced Bronchospasm
Brief Title: Study of Oglemilast for the Prevention of Asthma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: GRC-MD-01
Record Dates: First submitted 2006-05-04; First posted 2006-05-05 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Exercise-Induced Asthma
Keywords: oglemilast; asthma; exercise; prevention; prophylaxis
MeSH Terms: conditions — Asthma, Exercise-Induced; Asthma; Motor Activity | interventions — oglemilast

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Oglemilast (Experimental)
  Interventions: Drug: Oglemilast
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oglemilast — Oglemilast, 15mg once per day, oral administration
  Arms: Oglemilast
Drug: Placebo — Dose-marched placebo, once per day, oral administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether it is effective in the treatment of exercise-induced asthma and investigate the safety of oglemilast.

ELIGIBILITY:
Inclusion Criteria:

* stable mild asthma patients who exhibit at least a 20% decrease in FEV1 following exercise.

Exclusion Criteria:

* pulmonary disease other than asthma, psychiatric illness, active cardiac disease, high blood pressure, history of substance abuse, current smokers.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2006-05; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of oglemilast as compared to placebo in preventing exercise-induced asthma following 15 days of treatment.

SECONDARY OUTCOMES:
To evaluate the safety of oglemilast over 2 weeks as determined by adverse events, physical examinations, vital signs, electrocardiograms, and laboratory examinations.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Forest Investigative Site, Los Angeles, California
  - Forest Investigative Site, North Dartmouth, Massachusetts